CLINICAL TRIAL: NCT03495973
Title: Prospective Observational Study on Stelara Assessing Efficacy and Healthcare Resource Utilization in Crohn's Disease (PROSE)
Brief Title: Prospective Observational Study on Ustekinumab (Stelara) Assessing Efficacy and Healthcare Resource Utilization in Crohn's Disease
Acronym: PROSE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108430; CNTO1275CRD4006 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Crohn's Disease (CD): Participants with CD will be assessed for the effectiveness of ustekinumab in accordance with national guidelines and routine standard of care. Data will be prospectively collected with the aid of the Swedish inflammatory bowel disease (IBD) registry, SWIBREG and medical records of each participant. Data will also be collected retrospectively from SWIBREG and other databases including national databases such as the participant registry in which cases the national databases will be considered source data.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Participants that are initiated on treatment with ustekinumab and are registered in Swibreg will be recruited into the cohort. All aspects of treatment and clinical management of participants will be in accordance with local clinical practice and applicable local regulations, and at the discretion of the participating physician.

SUMMARY:
The main purpose of this study is to assess ustekinumab's ability to induce clinical response and remission ("effectiveness") at Week 16 and remission at Week 52 and Week 104 in participants with Crohn's disease (CD). Response and remission will be assessed using clinical parameters. Retention rate at week 52 and 104 will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of CD confirmed by investigator
* Participants with active CD who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a biologic therapy or have medical contraindications to such therapies
* The participant must sign informed consent before enrollment in the study. The consent form permits extraction of data from SWIBREG at baseline and during participation of the study and linkages to the Patient Registry (Patientregistret), SCB's registry USA for occupational details (Longitudinell integrationsdatabas for sjukforsakrings- och arbetsmarknadsstudi er), the Social Insurance registry on long-term sick leave (Forsakringskassans register gallande sjukskrivningar) and the Prescription registry (Lakemedelsregistret)
* The participant must have been initiated on treatment with ustekinumab within the last 2 weeks (that is including those who already discontinued) or started on ustekinumab treatment less than (<) 3 months ago if treatment start was documented in SWIBREG within 2 weeks of onset and has a record of Harvey Bradshaw Index (HBI) when starting ustekinumab

Exclusion Criteria:

* The participant is enrolled in a clinical trial (randomized or non-randomized) in which the treatment of CD is dictated by a study protocol. If the participant is participating in another observational study (non-interventional), the participant may be included in this observational study
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 60 days before the start of the study or the first data collection time point
* Participants who started ustekinumab despite contraindications for use
* Participants with planned stop of treatment with ustekinumab within 24 months from onset of treatment, that is bridging to other treatment or pregnancy planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed Crohn's disease (CD) aged over 18 years treated with ustekinumab.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-11-22 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 16, Based on Harvey Bradshaw Index (HBI) | Week 16
  Clinical response for Crohn's disease (CD) is assessed by Harvey Bradshaw Index (HBI) and is defined as decrease of 3 points in baseline HBI score. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 16, Based on HBI | Week 16
  Clinical remission for CD is assessed by HBI and is defined as HBI less than (<)5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score indicates: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 52, Based on HBI | Week 52
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 104, Based on HBI | Week 104
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 52 and 104, Based on HBI | Week 52 and 104
  Clinical response for CD is assessed by HBI and is defined as decrease of 3 points in baseline HBI score. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 52 and 104 who are Remitters at 16 Weeks | Week 52 and 104
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 104 who are Remitters at 52 Weeks | Week 104
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Percentage of Participants with Clinical Remission at Week 52 and 104 who are Responders at 16 Weeks | Week 52 and 104
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. Responders are defined as the participants with decrease of 3 points in baseline HBI score. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease.
Percentage of Participants in Clinical Remission Overtime | Up to Week 104
  Clinical remission for CD is assessed by HBI and is defined as HBI <5. HBI consists of clinical parameters: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicates more severe disease.
Percentage of Participants with Corticosteroid Free Remission at Week 52 and 104 | Week 52 and 104
  Participants on corticosteroids at baseline will be analyzed according to the percentage of participants in remission at week 52 and 104 without corticosteroids to assess corticosteroids free remission.
Participant's Time off Corticosteroids | Up to week 104
  Duration for which participants were off from corticosteroids will be determined.
Percentage of Participants in Every 12 weeks/8 weeks (q12 w/q8 w) maintenance groups at Week 16 | Week 16
  Percentage of participants in q12 w/q8 w maintenance groups will be determined at Week 16.
Percentage of Participants on Initial q12 w Maintenance Dose Escalated from q12 w to q8 w in Year 1 and 2 | Year 1 and 2
  Percentage of participants on initial q12 maintenance dose escalated from q12 w to q8 w in Year 1 and 2 will be determined.
Percentage of Participants with Dose Optimization | Year 1 and 2
  Percentage of participants with dose optimized to other dose than 90 milligram (mg) q8 w/q12 w in maintenance in Year 1 and 2 will be determined.
Average Maintenance Dose per Month | Week 52 and 104
  Average maintenance dose (in mg) taken per month will be determined.
Mean Change from Baseline in Fecal Calprotectin (fCal) Levels at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  Mean change from baseline in fCal (inflammatory biomarker) levels will be determined.
Mean Change from Baseline in C-reactive Protein (CRP) Levels at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  Mean change from baseline in C-reactive protein (CRP) (inflammatory biomarker) levels will be determined.
Percentage of Participants with fCal Less Than (<)250 milligram per kilogram (mg/kg) | Week 16, 52 and 104
  Percentage of participants with fCal <250 mg/kg will be determined.
Percentage of Participants with fCal levels <250 mg/kg at Week 16, 52 and 104 | Week 16, 52 and 104
  Percentage of participants with fCal levels <250 mg/kg at Week 16, 52 and 104 will be determined in total and amongst participants with fCal levels greater than (>)250 mg/kg at baseline.
Percentage of Participants with Normalization of Plasma-CRP (P-CRP) | Week 16, 52 and 104
  Percentage of participants with normalization of P-CRP in in participants with abnormal P-CRP at baseline will be reported. Normalization of P-CRP is defined as the high-sensitive (Hs)-CRP level <3 milligram per Liter (mg/L) or CRP below threshold of abnormal CRP concentration.
Change from Baseline in Short Health Scale (SHS) Score at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  Quality of life will be assessed by SHS score. SHS is a health related quality of life (HRQoL) questionnaire in which the participants rate the disease impact on 4 important aspects of subjective health (symptoms, function, worry, and general well-being). Responses are scored on 100-mm visual analogue scales and presented as individual scores for each of the four questions. The scores are then added for a total score. Total score ranges from 0 (low disease activity) to 100 (high disease activity).
Change from Baseline in EuroQoL 5-Dimension 5-Level Health Status (EQ-5D-5L) Questionnaire at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  Quality of life will be assessed by EQ-5D-5L score. The EQ-5D-5L descriptive system comprises following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of 5 dimension is divided into 5 levels of perceived problems (Level 1: no problem, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems, and Level 5: extreme problems). The participant selects an answer for each of 5 dimensions considering response that best matches his or her health "today". The descriptive system can be represented as a health state.
Change from Baseline in EQ-5D-5L Visual Analog Scale (VAS) at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  The EQ-VAS self-rating scale records respondent's own assessment of his or her overall health status at time of completion, on a scale of 0 (worst imaginable health) to 100 (best imaginable health).
Change from Baseline in the Presence of Extra Intestinal Manifestations at Week 16, 52 and 104 | Baseline, Week 16, 52 and 104
  Change in the presence of extra intestinal manifestations, that is arthralgia, peripheral arthritis, anchylosing spondylitis, uveitis, erythema nodosum, pyoderma gangrenosum, primary sclerosing cholangitis, psoriatic arthritis and psoriasis will be determined.
Healthcare Resource: Number of Imaging Procedures | Up to week 104
  Number of imaging procedures completed as a part of healthcare resources used in participants will be reported.
Healthcare Resource: Number of Laboratory Test | Up to Week 104
  Number of Laboratory tests completed as a part of healthcare resources used in participants will be reported.
Healthcare Resource: Number of Surgical Procedures | Up to Week 104
  Number of surgical procedures completed as a part of healthcare resources used in participants will be reported.
Healthcare Resource: Number of Dual Energy X-ray Absorptiometry (DEXA) Scans | Up to Week 104
  Number of DEXA scans performed as a part of healthcare resources used will be reported.
Healthcare Resource: Number of Participants with Endoscopies Performed | Up to Week 104
  Number of participants with endoscopies performed as a part of healthcare resources used will be reported.
Healthcare Resource: Number of Days of Hospitalization | Up to Week 104
  Number of days of hospitalization (defined as number of days from the day of admission to discharge) as a part of healthcare resources used will be reported.
Healthcare Resource: Number of Sick-Leaves | Up to Week 104
  Number of sick-leaves taken by participants as a part of healthcare resources used will be reported.
Healthcare Resource: Number of Participants Using Concomitant Treatment | Up to Week 104
  Number of participants using concomitant treatment as a part of healthcare resources used will be reported.
Healthcare Resource: Number of Health Care Visits | Up to Week 104
  Number of health care visits to nurses, dieticians and doctors as a part of healthcare resources used will be reported.
Number of Participants with Malignancy | Up to Week 104
  Number of participants with malignancy developed during the study will be reported.
Number of Participants Requiring Antibiotics for any Infection Occurred During the Study | Up to Week 104
  Number of participants requiring antibiotics for any infection occurred during the study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Universitetssjukhuset Orebro, Örebro, Sweden